CLINICAL TRIAL: NCT06198400
Title: Indocyanine Green Fluorescence in Evaluation of Post-resection Pancreatic Remnant Perfusion After Pancreaticoduodenectomy
Brief Title: Indocyanine Green Fluorescence in Evaluation of Pancreatic Remnant Perfusion.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Štěpán-Ota Schütz, Surgical resident, Postgraduate student, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MO1012
Record Dates: First submitted 2023-12-06; First posted 2024-01-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Fistula
Keywords: Pancreatic surgery; ICG; Minimal invasive surgery,; Pancreatic cancer; Pancreatic perfusion
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients undergoing the pancreaticoduodenectomy (Experimental): All consecutive patients undergoing the pancreaticoduodenectomy at our institution in the 1.5.2024-31.12.2026 period will be enrolled in this study.
  Interventions: Diagnostic Test: Perioperative assessment of the perfusion of post-resection pancreatic remnant using indocyanine green-VerDye

INTERVENTIONS:
Diagnostic Test: Perioperative assessment of the perfusion of post-resection pancreatic remnant using indocyanine green-VerDye — The adequacy of the vascular supply of the post resection pancreatic remnant after pancreatic neck division will be evaluated using ICG detector. Indocyanine green fluorescence product -Verdye™ will be intravenously applied. The application of the substance will be performed according to the current consensus statement and recommendation

SUMMARY:
Main goal of this study is to evaluate the blood flow in a post resection pancreatic remnant after pancreaticoduodenectomy with use of indocyanine green fluorescence. If the hypothesis will be proven, evaluation of perfusion of the pancreatic remnant with indocyanine green could be used to estimate the increased risk of the development of pancreatic fistula.

DETAILED DESCRIPTION:
Pancreatoduodenectomy is associated with nearly 25% incidence of postoperative complications. One of the most severe complications is a postoperative pancreatic fistula. The exact cause of postoperative fistula development is still unknown, but it appears to be multifactorial. Proper perfusion of pancreatic remnant is essential for the healing of pancreaticojejunostomy. To date, there is no method to reliably evaluate the vascular supply of the remnant. One of the methods for assessment of organ perfusion is the indocyanine green fluorescence. This study aims to determine if indocyanine green fluorescence is a reliable method to measure the perfusion of the post-resection pancreatic remnant. Secondary outcome is to determine, if perioperative evaluation of the vascular supply of the postresection remnant may predict the increased risk of the postoperative pancreatic fistula development.

This study is designed as a prospective experimental study. All consecutive patients undergoing open pancreaticoduodenectomy at our department in the 1.5.2024-31.12.2026 period will be enrolled. Exclusion criteria are allergy to indocyanine green and refusal by the patient.The adequacy of the vascular supply of the post-resection pancreatic remnant will be perioperatively evaluated using fluorescence detector. Patients will be divided into two groups. Those with hazardous and non-hazardous vascular supply. The incidence of pancreatic fistula in both groups is to be compared. Postoperative data including morbidity, mortality, hospital stay, intensive care unit stay and postoperative fistula development will be collected.

If a perioperative assessment of the perfusion of post-resection pancreatic remnant using indocyanine green is proven to be a suitable method to estimate the increased risk of the pancreatic fistula, the list of the existing known risk factors could be expanded. In the most high-risk patients the modification of the surgical procedure could be considered.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing open pancreaticoduodenectomy at our department in the selected period

Exclusion Criteria:

* Allergy to indocyanine green
* Refusal by the patient
* Mini-invasive procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the blood flow in pancreatic remnant with use of ICG | Intraoperatively: 5-10 minutes
  Primary outcome of this study is to evaluate the blood flow in a post resection pancreatic remnant after pancreaticoduodenectomy with use of ICG fluorescence.

SECONDARY OUTCOMES:
Correlation between ICG perfusion and development of pancreatic fistula | From admission to discharge, up to 2 weeks
  Secondary outcome of this study is to find possible correlation between ICG finding and higher rate of postoperative pancreatic fistula development which could lead to establishment of new predictive risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Radek Pohnán, Study Director — Department of Surgery, Second Faculty of Medicine of Charles University and Military University Hospital Prague, Czech Republic
Locations (1):
- Department of Surgery, Second Faculty of Medicine of Charles University and Military University Hospital Prague, Czech Republic, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Rawla P, Sunkara T, Gaduputi V. Epidemiology of Pancreatic Cancer: Global Trends, Etiology and Risk Factors. World J Oncol. 2019 Feb;10(1):10-27. doi: 10.14740/wjon1166. Epub 2019 Feb 26. PMID 30834048
- [Result] Karim SAM, Abdulla KS, Abdulkarim QH, Rahim FH. The outcomes and complications of pancreaticoduodenectomy (Whipple procedure): Cross sectional study. Int J Surg. 2018 Apr;52:383-387. doi: 10.1016/j.ijsu.2018.01.041. Epub 2018 Feb 10. PMID 29438817
- [Result] Rousek M, Whitley A, Kachlik D, Balko J, Zaruba P, Belbl M, Nikov A, Ryska M, Gurlich R, Pohnan R. The dorsal pancreatic artery: A meta-analysis with clinical correlations. Pancreatology. 2022 Mar;22(2):325-332. doi: 10.1016/j.pan.2022.02.002. Epub 2022 Feb 11. PMID 35177332
- [Result] Nahm CB, Connor SJ, Samra JS, Mittal A. Postoperative pancreatic fistula: a review of traditional and emerging concepts. Clin Exp Gastroenterol. 2018 Mar 15;11:105-118. doi: 10.2147/CEG.S120217. eCollection 2018. PMID 29588609
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Result] Bengtsson A, Andersson R, Ansari D. The actual 5-year survivors of pancreatic ductal adenocarcinoma based on real-world data. Sci Rep. 2020 Oct 2;10(1):16425. doi: 10.1038/s41598-020-73525-y. PMID 33009477
- [Result] de Muynck LDAN, White KP, Alseidi A, Bannone E, Boni L, Bouvet M, Falconi M, Fuchs HF, Ghadimi M, Gockel I, Hackert T, Ishizawa T, Kang CM, Kokudo N, Nickel F, Partelli S, Rangelova E, Swijnenburg RJ, Dip F, Rosenthal RJ, Vahrmeijer AL, Mieog JSD. Consensus Statement on the Use of Near-Infrared Fluorescence Imaging during Pancreatic Cancer Surgery Based on a Delphi Study: Surgeons' Perspectives on Current Use and Future Recommendations. Cancers (Basel). 2023 Jan 20;15(3):652. doi: 10.3390/cancers15030652. PMID 36765609
- [Result] Strasberg SM, Drebin JA, Mokadam NA, Green DW, Jones KL, Ehlers JP, Linehan D. Prospective trial of a blood supply-based technique of pancreaticojejunostomy: effect on anastomotic failure in the Whipple procedure. J Am Coll Surg. 2002 Jun;194(6):746-58; discussion 759-60. doi: 10.1016/s1072-7515(02)01202-4. PMID 12081065
- [Result] Boni L, David G, Mangano A, Dionigi G, Rausei S, Spampatti S, Cassinotti E, Fingerhut A. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. Surg Endosc. 2015 Jul;29(7):2046-55. doi: 10.1007/s00464-014-3895-x. Epub 2014 Oct 11. PMID 25303914
- [Result] CHERRICK GR, STEIN SW, LEEVY CM, DAVIDSON CS. Indocyanine green: observations on its physical properties, plasma decay, and hepatic extraction. J Clin Invest. 1960 Apr;39(4):592-600. doi: 10.1172/JCI104072. No abstract available. PMID 13809697
- [Result] Keller DS, Ishizawa T, Cohen R, Chand M. Indocyanine green fluorescence imaging in colorectal surgery: overview, applications, and future directions. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):757-766. doi: 10.1016/S2468-1253(17)30216-9. PMID 28895551
- [Result] Hackethal A, Hirschburger M, Eicker SO, Mucke T, Lindner C, Buchweitz O. Role of Indocyanine Green in Fluorescence Imaging with Near-Infrared Light to Identify Sentinel Lymph Nodes, Lymphatic Vessels and Pathways Prior to Surgery - A Critical Evaluation of Options. Geburtshilfe Frauenheilkd. 2018 Jan;78(1):54-62. doi: 10.1055/s-0043-123937. Epub 2018 Jan 22. PMID 29375146
- [Result] Degett TH, Andersen HS, Gogenur I. Indocyanine green fluorescence angiography for intraoperative assessment of gastrointestinal anastomotic perfusion: a systematic review of clinical trials. Langenbecks Arch Surg. 2016 Sep;401(6):767-75. doi: 10.1007/s00423-016-1400-9. Epub 2016 Mar 11. PMID 26968863
- [Result] Doussot A, Decrock M, Calame P, Georges P, Turco C, Lakkis Z, Heyd B. Fluorescence-based pancreas stump perfusion is associated with postoperative acute pancreatitis after pancreatoduodenectomy a prospective cohort study. Pancreatology. 2021 Sep;21(6):1023-1029. doi: 10.1016/j.pan.2021.05.009. Epub 2021 May 18. PMID 34030965
- [Result] Marchegiani G, Perri G, Burelli A, Zoccatelli F, Andrianello S, Luchini C, Donadello K, Bassi C, Salvia R. High-risk Pancreatic Anastomosis Versus Total Pancreatectomy After Pancreatoduodenectomy: Postoperative Outcomes and Quality of Life Analysis. Ann Surg. 2022 Dec 1;276(6):e905-e913. doi: 10.1097/SLA.0000000000004840. Epub 2021 Mar 4. PMID 33914471
- [Result] Baiocchi GL, Diana M, Boni L. Indocyanine green-based fluorescence imaging in visceral and hepatobiliary and pancreatic surgery: State of the art and future directions. World J Gastroenterol. 2018 Jul 21;24(27):2921-2930. doi: 10.3748/wjg.v24.i27.2921. PMID 30038461
- [Result] Hu BY, Wan T, Zhang WZ, Dong JH. Risk factors for postoperative pancreatic fistula: Analysis of 539 successive cases of pancreaticoduodenectomy. World J Gastroenterol. 2016 Sep 14;22(34):7797-805. doi: 10.3748/wjg.v22.i34.7797. PMID 27678363
- [Result] Fuks D, Piessen G, Huet E, Tavernier M, Zerbib P, Michot F, Scotte M, Triboulet JP, Mariette C, Chiche L, Salame E, Segol P, Pruvot FR, Mauvais F, Roman H, Verhaeghe P, Regimbeau JM. Life-threatening postoperative pancreatic fistula (grade C) after pancreaticoduodenectomy: incidence, prognosis, and risk factors. Am J Surg. 2009 Jun;197(6):702-9. doi: 10.1016/j.amjsurg.2008.03.004. Epub 2008 Sep 7. PMID 18778804
- [Result] Gaujoux S, Cortes A, Couvelard A, Noullet S, Clavel L, Rebours V, Levy P, Sauvanet A, Ruszniewski P, Belghiti J. Fatty pancreas and increased body mass index are risk factors of pancreatic fistula after pancreaticoduodenectomy. Surgery. 2010 Jul;148(1):15-23. doi: 10.1016/j.surg.2009.12.005. PMID 20138325
- [Result] Pedrazzoli S. Pancreatoduodenectomy (PD) and postoperative pancreatic fistula (POPF): A systematic review and analysis of the POPF-related mortality rate in 60,739 patients retrieved from the English literature published between 1990 and 2015. Medicine (Baltimore). 2017 May;96(19):e6858. doi: 10.1097/MD.0000000000006858. PMID 28489778
- [Derived] Schutz SO, Rousek M, Zaruba P, Husarova T, Pohnan R. Indocyanine green fluorescence in the evaluation of post-resection pancreatic remnant perfusion after a pancreaticoduodenectomy: a clinical study protocol. BMC Surg. 2024 Sep 14;24(1):261. doi: 10.1186/s12893-024-02559-0. PMID 39272087
- See also: Indocyanine Green-Fluorescent Pancreatic Perfusion-Guided Resection of Distal Pancreas in Solid Pseudopapillary Neoplasm: Usefulness and Feasibility During Pancreaticobiliary Surgery — https://www.e-jmis.org/journal/view.html?doi=10.7602/jmis.2018.21.1.43